CLINICAL TRIAL: NCT00886171
Title: Effects of Social Skills and Physical Activity Training on Recreational Activities in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Sarah-Jeanne Salvy, Assistant Professor, University at Buffalo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB#2175
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Social Skills; Physical Activity
Keywords: social skills; physical activity; peer relationships; childhood obesity; changes in physical activity; changes in social involvement
MeSH Terms: conditions — Social Skills; Motor Activity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Skills Training (Experimental)
  Interventions: Behavioral: Social Skills Training
- Physical Activity Training (Experimental)
  Interventions: Behavioral: Physical Activity Training

INTERVENTIONS:
Behavioral: Social Skills Training — Social skills group will consist of one session (60 minutes) per week for 8 weeks
  Arms: Social Skills Training
Behavioral: Physical Activity Training — Physical activity groups consist of one session (60 minutes) per week for 8 weeks
  Arms: Physical Activity Training

SUMMARY:
The purpose of this study is to examine the effect of social skills training on adolescents physical activity levels. For one week at the beginning and end of the study teens will wear a BioTrainer to measure their activity levels and also wear a pager to communicate the types of activities they are doing throughout the day. For 8 weeks participants will be randomized into one of two groups, a social skills training group or a physical activity group.

The investigators predict that both groups will experience an increase in physical activity and social involvement (decrease time spent alone).

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 12-14
* Youth who encounter problematic relationships with their peers

Exclusion Criteria:

* Youth should have no psychopathology, developmental disabilities, or asthma that would limit participation
* Youth should have no cold or upper respiratory distress or a condition that could influence their activities
* Youth should not be taking medications that could affect their level of activity

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
physical activity levels | pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Salvy, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Division of Behavioral Medicine, Buffalo, New York, United States